CLINICAL TRIAL: NCT02580331
Title: 1% Metformin Gel as Local Drug Delivery in the Treatment of Class II Furcation Defects: A Randomized Controlled Clinical Trial
Brief Title: 1% Metformin Gel in the Treatment of Class II Furcation Defects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor, Government Dental College and Research Institute, Bangalore, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2013-2014S
Record Dates: First submitted 2015-10-18; First posted 2015-10-20 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SRP and placebo (Placebo Comparator): Oral prophylaxis followed by placement of placebo gel
  Interventions: Drug: SRP and placebo
- SRP and 1% metformin (Active Comparator): Oral prophylaxis followed by placement of 1% metformin gel
  Interventions: Drug: SRP and 1% metformin

INTERVENTIONS:
Drug: SRP and placebo — Placement of placebo gel into classII furcation defects after scaling and root planing
  Other Names: Group 1
  Arms: SRP and placebo
Drug: SRP and 1% metformin — Placement of 1% metformin gel into classII furcation defects after scaling and root planing
  Other Names: Group 2
  Arms: SRP and 1% metformin

SUMMARY:
Metformin (MF), a biguanide group of anti-diabetic drug has been shown to enhance osteoblasts differentiation and inhibit osteoclast differentiation in vitro, thus may exhibit a favourable effect on alveolar bone. The present study aims to explore the efficacy of 1% MF gel as a local drug delivery system in adjunct to scaling and root planing (SRP) for the treatment of Class II furcation defects in comparison with placebo gel.

DETAILED DESCRIPTION:
Background: Metformin (MF), a biguanide group of anti-diabetic drug has been shown to enhance osteoblasts differentiation and inhibit osteoclast differentiation in vitro, thus may exhibit a favourable effect on alveolar bone. The present study aims to explore the efficacy of 1% MF gel as a local drug delivery system in adjunct to scaling and root planing (SRP) for the treatment of Class II furcation defects in comparison with placebo gel.

Methods: Sixty four patients with single mandibular buccal class II furcation defects were categorized into two treatment groups: SRP plus 1% MF (group 1) and SRP plus placebo (group 2). Clinical parameters were recorded at baseline, 3 months, 6 months, and 9 months, and radiographic parameters were recorded at baseline, 6 months, and 9 months. Defect fill at baseline, 6 months, and 9 months was calculated on standardized radiographs using image analysis software.

ELIGIBILITY:
Inclusion Criteria:

1. the presence of buccal Class II furcation defects in endodontically vital, asymptomatic mandibular first molars with a radiolucency in the furcation area on an intraoral periapical radiograph with PD≥ 5 mm and horizontal PD≥3 mm following phase I therapy (SRP)

Exclusion Criteria:

* patients with known systemic disease; patients with known or suspected allergy to the MF; patients receiving systemic MF therapy; patients with aggressive periodontitis; patients using tobacco in any form; patients with alcoholism; patients who were immunocompromised; pregnant or lactating females.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2014-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Bone defect fill | baseline to 9 months
  Assesed in percentage

SECONDARY OUTCOMES:
modified sulcus bleeding index | baseline to 9 months
  scale 0-3
plaque index | baseline to 9 months
  scale 0-3
pocket probing depth | baseline to 9 months
  measured in mm
relative vertical clinical attachment level | baseline to 9 months
  measured in mm
relative horizontal clinical attachment level | baseline to 9 months
  measured in mm

CONTACTS AND LOCATIONS:
Overall Officials: A R Pradeep, MDS, Principal Investigator — GDCRI
Locations (1):
- Government Dental College and Research Institute, Bangalore, Karnataka, India